CLINICAL TRIAL: NCT07026227
Title: Clinical Study on the Effect of Xuebijing in Alleviating Acute Kidney Injury After High-voltage Electrical Burns by Inhibiting Neutrophils, Inflammatory Cells, and Reactive Oxygen Species
Brief Title: Effect of Xuebijing in Alleviating Acute Kidney Injury After High-voltage Electrical Burns
Acronym: Xuebijing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, Xin Xue, Principal Investigator, The First Hospital of Hebei Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S-00312
Record Dates: First submitted 2025-06-04; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Acute Kidney Injury
Keywords: Acute Kidney Injury; Xuebijing; neutrophils; inflammatory cells
MeSH Terms: conditions — Acute Kidney Injury | interventions — Xuebijing

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Xuebijing + Conventional Treatment) (Experimental): Participants randomized to this arm received conventional treatment for acute kidney injury (AKI) following high-voltage electrical burns, plus Xuebijing injection.
  Interventions: Drug: Xuebijing Injection
- Control Group (Conventional Treatment Only) (Active Comparator): Participants randomized to this arm received conventional treatment alone for acute kidney injury (AKI) following high-voltage electrical burns.
  Interventions: Procedure: Conventional Treatment for High-Voltage Electrical Burns and AKI

INTERVENTIONS:
Drug: Xuebijing Injection — Xuebijing injection (Tianjin Hongri Pharmaceutical Co., Ltd., National Drug Standard Z20040033).
  Arms: Study Group (Xuebijing + Conventional Treatment)
Procedure: Conventional Treatment for High-Voltage Electrical Burns and AKI — Standard multidisciplinary care including general burn assessment, wound management (cleaning, debridement, dressings), fluid resuscitation as per burn protocols, management of electrolyte imbalances
  Arms: Control Group (Conventional Treatment Only)

SUMMARY:
High-voltage electrical burns frequently lead to acute kidney injury (AKI), a severe complication with high mortality. This study investigated the clinical efficacy and safety of Xuebijing injection, a traditional Chinese medicine preparation, in alleviating AKI in patients with high-voltage electrical burns. The study hypothesized that Xuebijing could improve renal outcomes by inhibiting neutrophils, inflammatory cells, and modulating reactive oxygen species (ROS).

This was a randomized, open-label, controlled clinical trial conducted at the Third Hospital of Hebei Medical University. Ninety-six adult patients admitted between February 2023 and December 2024 with AKI secondary to high-voltage electrical burns (burn area >30% TBSA or third-degree burns >10% TBSA, meeting AKI diagnostic criteria) were enrolled. Patients were randomized (1:1) into two groups: a study group (n=48) receiving conventional treatment plus Xuebijing injection (50 mL diluted in 100 mL 0.9% sodium chloride, IV drip, twice daily for 7 days), and a control group (n=48) receiving conventional treatment alone. Laboratory personnel assessing outcomes were blinded to group allocation where feasible.

Primary outcomes included changes in kidney function markers (Blood Urea Nitrogen [BUN], Serum Creatinine [SCr], 24-hour urinary protein), inflammatory markers (neutrophils, C-reactive protein [CRP], Interleukin-18 [IL-18], Interleukin-6 [IL-6]), and oxidative stress markers (Superoxide Dismutase [SOD], Malondialdehyde [MDA]). These were measured at baseline (1 hour before treatment) and 7 days post-treatment. Adverse reactions were also monitored.

ELIGIBILITY:
Inclusion Criteria:

1. Burns caused by high-voltage electrical injury, with a serum creatinine (Cr) level increase of at least 26.5 μmol/L within 48 hours, or urine output less than 0.5 mL/(kg•h) sustained for 6 hours, or a Cr level rising to 1.5 times the baseline within 7 days.
2. Burn area greater than 30% of the total body surface area (TBSA), or third-degree burns covering more than 10% of the TBSA.
3. All patients were admitted within 24 hours of the burn injury and survived for at least 14 days post-admission.
4. All patients were aged ≥18 years.

Exclusion Criteria:

1. Radiation exposure or nephrotoxic drug exposure within 5 days prior to admission.
2. Pre-existing AKI at any stage, according to KDIGO criteria.
3. Chronic kidney disease for any reason, with a glomerular filtration rate (GFR) ≤ 60 mL/(min•1.73 m²) for at least 3 months.
4. Post-kidney transplant patients.
5. Patients who had received or required continuous renal replacement therapy (CRRT) within 7 days.
6. Anuria (urine output <100 mL/d) preventing sample collection.
7. Patients with malignant tumors.
8. Patients with autoimmune diseases requiring long-term steroid therapy.
9. Patients who had received high-dose steroid treatment within the past month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2023-08-20 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Change in Serum Creatinine (SCr) Level | Baseline (1 hour before treatment initiation) and 7 days after treatment initiation.
  Change in serum creatinine concentration from baseline to 7 days post-treatment. SCr is a key marker for assessing kidney function and injury. Measured in μmol/L.
Change in Blood Urea Nitrogen (BUN) Level | Baseline (1 hour before treatment initiation) and 7 days after treatment initiation.
  Change in blood urea nitrogen concentration from baseline to 7 days post-treatment. BUN is another important marker for assessing kidney function. Measured in mmol/L.
Change in 24-hour Urinary Protein Level | Baseline (1 hour before treatment initiation, based on a 24-hour collection prior) and 7 days after treatment initiation (based on a 24-hour collection ending on day 7).
  Change in the amount of protein excreted in urine over a 24-hour period from baseline to 7 days post-treatment. This indicates the extent of glomerular and tubular damage. Measured in mg/24h.

SECONDARY OUTCOMES:
Change in Neutrophil Count | Baseline (1 hour before treatment initiation) and 7 days after treatment initiation.
  Change in peripheral blood neutrophil count from baseline to 7 days post-treatment. Neutrophils are key inflammatory cells involved in AKI pathogenesis. Measured in 10^9/L.
Change in C-Reactive Protein (CRP) Level | Baseline (1 hour before treatment initiation) and 7 days after treatment initiation.
  Change in serum C-reactive protein concentration from baseline to 7 days post-treatment. CRP is a systemic marker of inflammation. Measured in mg/L.
Change in Interleukin-18 (IL-18) Level | Baseline (1 hour before treatment initiation) and 7 days after treatment initiation.
  Change in serum Interleukin-18 concentration from baseline to 7 days post-treatment. IL-18 is a pro-inflammatory cytokine implicated in kidney injury. Measured in ng/mL (or pg/mL, check units from actual lab).
Change in Interleukin-6 (IL-6) Level | Baseline (1 hour before treatment initiation) and 7 days after treatment initiation.
  Change in serum Interleukin-6 concentration from baseline to 7 days post-treatment. IL-6 is another key pro-inflammatory cytokine. Measured in ng/mL (or pg/mL, check units from actual lab).
Change in Superoxide Dismutase (SOD) Level | Baseline (1 hour before treatment initiation) and 7 days after treatment initiation.
  Change in serum Superoxide Dismutase activity from baseline to 7 days post-treatment. SOD is an antioxidant enzyme. Measured in U/mL.
Change in Malondialdehyde (MDA) Level | Baseline (1 hour before treatment initiation) and 7 days after treatment initiation.
  Change in serum Malondialdehyde concentration from baseline to 7 days post-treatment. MDA is a marker of lipid peroxidation and oxidative stress. Measured in nmol/mL.
Incidence of Adverse Reactions | Throughout the 7-day treatment period.
  Number and type of adverse reactions (e.g., skin rashes, nausea, fever, abdominal pain, etc.) reported by participants or observed by investigators in each group during the 7-day treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Yinghui Pang, BSN, Principal Investigator — First Hospital of Hebei Medical University
Locations (1):
- First Hospital of Hebei Medical University, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] He X, Li N, Ma L, Yang M, Ren L, Hao J, Xue X, Pang Y. Xuebijing alleviates high-voltage electrical burn-induced acute kidney injury by inhibiting neutrophils and inflammation. Sci Rep. 2025 Aug 19;15(1):30410. doi: 10.1038/s41598-025-11977-w. PMID 40830157